CLINICAL TRIAL: NCT00035906
Title: Research Study in Patients With Persistent Macular Edema Due to Diabetic Retinopathy, Retinal Vein Occlusion, Uveitis, or Irvine-Gass Syndrome
Brief Title: Research Study in Patients With Persistent Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: Oculex Pharmaceuticals (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: DC-103-06-03
Record Dates: First submitted 2002-05-06; First posted 2002-05-07 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Diabetes; Macular Edema; Diabetic Retinopathy; Retinal Disease; Uveitis, Posterior
Keywords: Diabetes; Macular Edema; Diabetic Macular Edema; Diabetic Retinopathy; Cystoid Macular Edema; Uveitis; Vision; Eye; Retina; Retinal Vein Occlusion; Irvine-Gass Syndrome
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema; Diabetic Retinopathy; Retinal Diseases; Uveitis, Posterior; Uveitis; Retinal Vein Occlusion

INTERVENTIONS:
Drug: DEX PS DDS®

SUMMARY:
The purpose of this clinical research study is to evaluate the safety and effectiveness of an investigational medication to treat macular edema that persists despite current treatment methods. Participants will be evaluated for improvement in vision and side effects.

Macular edema is a condition that affects the back of the eye (retina). It frequently occurs in people who have a history of diabetes, and is also associated with high blood pressure, uveitis, and previous eye surgery. The main symptom of macular edema is decreased vision, generally a blurring of central vision.

There are no direct costs to participants for assessments and treatment as defined in the study protocol. All candidates must be available for required scheduled visits during the trial's 6-month follow-up period. Although the disease called age-related macular degeneration (AMD) affects the same region of the eye as macular edema, they are not the same condition and AMD is not studied in this research trial.

ELIGIBILITY:
Inclusion: Persistent macular edema associated with diabetic retinopathy, uveitis, retinal vein occlusion, or Irvine-Gass syndrome, persisting at least 90 days after laser treatment or medical management by a physician.

Exclusion: Females who are pregnant or lactating, and females of childbearing potential not using adequate birth control for the duration of the study. Any intraocular procedures or laser treatment less than 90 days before enrollment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2001-10; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oculex Pharmaceuticals, Sunnyvale, California, United States

REFERENCES:
- [Derived] Haller JA, Kuppermann BD, Blumenkranz MS, Williams GA, Weinberg DV, Chou C, Whitcup SM; Dexamethasone DDS Phase II Study Group. Randomized controlled trial of an intravitreous dexamethasone drug delivery system in patients with diabetic macular edema. Arch Ophthalmol. 2010 Mar;128(3):289-96. doi: 10.1001/archophthalmol.2010.21. PMID 20212197
- [Derived] Kuppermann BD, Chou C, Weinberg DV, Whitcup SM, Haller JA, Blumenkranz MS; Dexamethasone DDS Phase II Study Group. Intravitreous dexamethasone effects on different patterns of diabetic macular edema. Arch Ophthalmol. 2010 May;128(5):642-3. doi: 10.1001/archophthalmol.2010.44. Epub 2010 Mar 8. No abstract available. PMID 20212194
- [Derived] Williams GA, Haller JA, Kuppermann BD, Blumenkranz MS, Weinberg DV, Chou C, Whitcup SM; Dexamethasone DDS Phase II Study Group. Dexamethasone posterior-segment drug delivery system in the treatment of macular edema resulting from uveitis or Irvine-Gass syndrome. Am J Ophthalmol. 2009 Jun;147(6):1048-54, 1054.e1-2. doi: 10.1016/j.ajo.2008.12.033. Epub 2009 Mar 9. PMID 19268890
- [Derived] Kuppermann BD, Blumenkranz MS, Haller JA, Williams GA, Weinberg DV, Chou C, Whitcup SM; Dexamethasone DDS Phase II Study Group. Randomized controlled study of an intravitreous dexamethasone drug delivery system in patients with persistent macular edema. Arch Ophthalmol. 2007 Mar;125(3):309-17. doi: 10.1001/archopht.125.3.309. PMID 17353400